CLINICAL TRIAL: NCT05257798
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY OPEN, PLACEBO CONTROLLED, STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY FOLLOWING A SINGLE DOSE OF PF-06823859 IN HEALTHY CHINESE PARTICIPANTS
Brief Title: A Study to Learn About The Study Medicine (Called PF-06823859) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: C0251007
Record Dates: First submitted 2022-02-03; First posted 2022-02-25 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PF-06823859 (Experimental): Participants will receive 900 mg of PF-06823859 via intravaneous (IV).
  Interventions: Drug: IFN-β inhibitor treatment
- Placebo (Placebo Comparator): Participants will receive placebo via IV.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IFN-β inhibitor treatment — PF-06823859 (IFN-β inhibitor) 100 mg/mL solution for injection
  Arms: PF-06823859
Other: Placebo — Placebo for PF-06823859, 0 mg/mL solution for injection
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to learn if the study medicine (called PF-06823859) is safe and how it is processed in healthy Chinese participants. This study is seeking participants who:

* Are between 18 to 45 years of age, inclusive, at the time of signing the Informed Consent Document (ICD).
* Are Chinese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12 lead ECG (electrocardiogram).
* Have a BMI (body mass index) of 19 to 27 kg/m2 (inclusive); and a total body weight >50 kg (110 lb).

All participants in this study will receive PF-06823859 or a placebo. A placebo does not have any medicine in it but looks just like the medicine being studied. PF-06823859 will be given as an infusion directly into a vein. We will compare the experiences of people receiving PF-06823859 to those of people who do not. This will help us determine if PF-06823859 is safe and how it behaves inside the human body.

Participants will take part in this study for up to 157 days. During this time, they will receive PF-06823859 or placebo and be observed for any effects.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double blind, sponsor open, placebo controlled study to evaluate the PK, safety, and tolerability following a single dose of PF 06823859 (900 mg) in healthy Chinese participants.

ELIGIBILITY:
1.1. Inclusion Criteria

1. Male and female participants must be 18 to 45 years of age, inclusive, at the time of signing the ICD (informed consent document).
2. Male and female Chinese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12 lead ECG (electrocardiogram).
3. BMI (body mass index) of 19 to 27 kg/m2 (inclusive); and a total body weight >50 kg (110 lb).

1.2. Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
2. History of HIV (human immunodeficiency virus) infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg (hepatitis B surface antigen), or HCVAb (hepatitis C antibody).
3. History of autoimmune disorders.
4. History of allergic or anaphylactic reaction to a therapeutic drug.
5. History of recent active infections within 28 days prior to the screening visit.
6. Participants with a fever within 7 days prior to dosing.
7. Infected with Mycobacterium TB (tuberculosis)
8. Contact with positive case of COVID (coronavirus disease)-19 or travel to an area defined as high risk by relevant authority in the past 14 days.
9. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
10. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
11. Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 83 participants screened in the study, among whom, 18 participants were assigned to the study treatments.
Groups:
- PF-06823859 900mg: Participants received a single intravenous (IV) infusion of PF-06823859 900 mg on Study Day 1
- Placebo: Participants received a single IV infusion of placebo on Study Day 1
Period: Treatment Phase
Arm/Group | PF-06823859 900mg | Placebo
Started | 15 | 3
Completed | 15 | 3
Not Completed | 0 | 0
Period: Follow-up Phase
Arm/Group | PF-06823859 900mg | Placebo
Started | 15 | 3
Completed | 14 | 3
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06823859 900mg | Placebo | Total
Number analyzed (Participants) | 15 | 3 | 18
Age, Continuous [Median (Full Range); unit: years] | 33.00 [21 to 41] | 28.00 [26 to 32] | 30.50 [21 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 13 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 15 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration(Cmax) for PF-06823859
Description: The Cmax was observed directly from data.
Time Frame: Days 1 (pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: The PK parameter analysis population included all randomized participants who received at least 1 dose of study intervention and at least 1 of the PK parameters was calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/mL)
Groups:
- PF-06823859 900 mg: Participants received a single intravenous (IV) infusion of PF-06823859 900 mg on Study Day 1
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
micrograms/milliliter (ug/mL) | 307.4 (17)

2. Primary Outcome: Time at Which Cmax Occured (Tmax) for PF-06823859 in Serum
Description: The Tmax was the time at which Cmax occurs
Time Frame: Days 1 (pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
hour (hr) | 1.52 [1.00 to 12.0]

3. Primary Outcome: Area Under the Concentration-time Profile From Time Zero to 14 Days (336 Hours) Post-dose (AUC14day) for PF-06823859 in Serum
Description: The AUC14day was area under the concentration-time profile from time zero to 14 days post-dose (336 hours)
Time Frame: Days 1 (pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
ug*hr/mL | 48550 (16)

4. Primary Outcome: Area Under the Concentration-time Profile From Time Zero to 28 Days (672 Hours) Post-dose (AUC28day) for PF-06823859 in Serum
Description: The AUC28day was area under the concentration-time profile from time zero to 28 days post-dose (672 hours)
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
ug*hr/mL | 73240 (17)

5. Primary Outcome: Area Under the Serum Concentration-time Profile From Time Zero Extrapolated to Infinite Time(AUCinf) for PF-06823859 in Serum.
Description: The AUCinf was area under the serum concentration-time profile from time zero extrapolated to infinite time
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
ug*hr/mL | 127100 (23)

6. Primary Outcome: Terminal Half-life (t1/2) for PF-06823859 in Serum.
Description: The t1/2 was terminal half-life (time required for the plasma concentration to decline by 50%).
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention and at least 1 of the PK parameters was calculated.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
day | 26.96 (2.6945)

7. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; or other serious situations such as important medical events. TEAEs were events between first dose of study drug and up to follow-up visit that were absent before treatment or that worsened after treatment. AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: From first dose of study drug/Day 1 to Day 157
Population: The safety analysis population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 15 | 3
Participants
  Participants with TEAEs | 14 | 2
  Participants with serious TEAEs | 0 | 0

8. Primary Outcome: Number of Participants With Pre-Specified Categorization for Vital Signs (Diastolic Blood Pressure)
Description: Vital signs measurements included supine blood pressure, diastolic blood pressure, pulse rate and temperature. For diastolic blood pressure, the reporting criteria is increase or decrease from baseline of >= 20mmHg or absolute value < 50 mmHg.
Time Frame: Days 1 (pre-dose),5,29,57,100,127 and 157.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 15 | 3
Participants | 1 | 0

9. Primary Outcome: Number of Participants With Pre-Specified Categorization for Vital Signs (Systolic Blood Pressure)
Description: Vital signs measurements included supine blood pressure, diastolic blood pressure, pulse rate and temperature. For systolic blood pressure, the reporting criteria is increase or decrease from baseline of >= 30 mm Hg or absolute value of <90 mmHg
Time Frame: Days 1 (pre-dose),5,29,57,100,127 and 157.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 15 | 3
Participants
  Systolic Blood Pressure (mmHg) Change >= 30 mmHg increase | 1 | 0
  Systolic Blood Pressure (mmHg) Change >= 30 mmHg decrease | 1 | 0

10. Primary Outcome: Number of Participants With Pre-Specified Categorization (Maximum Change From Baseline) for ECG Data
Description: Standard 12 lead ECGs utilizing limb leads (with a 10 second rhythm strip) were collected at pre-specified times using an ECG machine that automatically calculates the heart rate and measures PR, QT, and QTc intervals and QRS complex. For Safely QTc assessments, absolute value of >450msec and < 480msec is defined as mild prolongation; absolute value between 480-500msec or an increase from baseline of 30 -60msec are defined as moderate prolongation; an absolute value of > 500msec or increase from baseline of >60 msec are defined as severe prolongation.
Time Frame: Days -1, 5,29,57,100,127 and 157.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 15 | 3
Participants | 0 | 0

11. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality).
Description: Safety laboratory assessments included urinalysis, hematology, chemistry and other. All the safety laboratory samples were collected following at least a 4-hour fast.
Time Frame: Days -1, 2, 5,8,15,29,57,100,127 and 157.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 15 | 3
Participants
  Ery. Mean Corpuscular HGB Concentration (g/L) < 0.9 ✖ Lower Limit Normal (LLN) | 1 | 0
  Lymphocytes (10^9/L) > 1.2 ✖ Upper Limit Normal (ULN) | 1 | 0
  Basophils (10^9/L) > 1.2 ✖ ULN | 1 | 0
  Eosinophils (10^9/L) > 1.2 ✖ ULN | 1 | 0
  Prothrombin Time (s) > 1.1 ✖ ULN | 1 | 0
  Bilirubin (micromol/L) > 1.5 ✖ ULN | 1 | 0
  Urate (mmol/L) > 1.2 ✖ ULN | 1 | 0
  pH (Scalar) >8 | 1 | 0
  URINE Erythrocytes (Scalar) >= 20 | 2 | 0
  URINE Leukocytes (Scalar) >= 20 | 2 | 0
  Ketones >= 1 | 1 | 0
  URINE Hemoglobin >= 1 | 2 | 0

12. Primary Outcome: Number of Participants With Viral Infections
Description: Viral infections surveillance was conducted throughout the study for cytomegalovirus (CMV), Epstein Barr virus (EBV), herpes simplex virus type 1 (HSV-1),herpes simplex virus type 2 (HSV-2), varicella zoster virus (VZV)， Human Herpes Virus 6 (HHV6) and COVID-19.
Time Frame: From Screening up to Day157
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 15 | 3
Participants | 3 | 0

13. Secondary Outcome: Area Under the Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (Clast) (AUClast) for PF-06823859 in Serum
Description: The AUClast was area under the serum concentration-time profile from time zero to the time of the last quantifiable concentration (Clast)
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
ug*hr/mL | 124700 (23)

14. Secondary Outcome: Clearance(CL) for PF-06823859 in Serum
Description: The CL was clearance.
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
L/hr | 0.007084 (23)

15. Secondary Outcome: Volume of Distribution at Steady State (Vss) for PF-06823859 in Serum
Description: The Vss was volume of distribution.
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
L | 5.800 (18)

16. Secondary Outcome: Mean Residence Time (MRT) for PF-06823859 in Serum
Description: The MRT was mean residence time.
Time Frame: Days 1(pre-dose, 1, 2, 6, 12 hours post dose), 2,3,5,15,29,43,57,71,100,127 and 157.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 10
Day | 34.13 (17)

17. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) of PF-06823859
Description: The percentage of participants with positive ADA was summarized.
Time Frame: Days 1 (pre-dose), 15,29, 57, 71, 100, 127 and 157.
Population: The immunogenicity analysis population included all randomized participants who received at least 1 dose of study intervention with at least 1 post-treatment anti-drug antibody determination.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 900 mg
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: From screening up to Day 157
Description: Serious adverse events(SAE) and non-serious AEs were recorded on the case report form.
Arm/Group | PF-06823859 900mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/3
Other Adverse Events (participants affected / at risk) | 14/15 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06823859 900mg (N=15) | Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0
Ear infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Urinary occult blood positive (Investigations) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT05257798/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT05257798/SAP_001.pdf